CLINICAL TRIAL: NCT07181967
Title: Evaluation of Streptococcus Mutans Reduction by Silver Diamine Fluoride vs. Fluoride Varnish: A Split-Mouth Study in Children
Brief Title: SDF vs Fluoride Varnish for Streptococcus Mutans Reduction in Children
Acronym: Streptococcus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ِAhmed kamel Abdel Naser soliman, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 17-2025-00013; 17-2025-00013 (Other Grant/Funding Number: Assuit university)
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries
Keywords: Silver Diamine Fluoride; Fluoride Varnish; Streptococcus mutans; Dental Plaque
MeSH Terms: conditions — Dental Caries; Dental Plaque | interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized controlled trial. Each child receives 38% silver diamine fluoride (SDF) on one side and 5% sodium fluoride varnish (FV) on the contralateral side. This within-subject design minimizes inter-individual variability, with each participant serving as their own control.
Who Masked: Outcomes Assessor
Masking Description: The operator and participants could not be blinded because 38% silver diamine fluoride (SDF) produces visible black staining of carious lesions. The outcome assessor for Streptococcus mutans (Dentocult SM test) was blinded; plaque samples were coded, and the assessor had no knowledge of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Diamine Fluoride (SDF) (Experimental): Application of 38% silver diamine fluoride (44,800 ppm F) to all eligible dentin caries lesions on the assigned side of the mouth. Single application per manufacturer's instructions.
  Interventions: Drug: Silver Diamine Fluoride (38%)
- Fluoride Varnish (FV) (Active Comparator): Application of 5% sodium fluoride varnish (22,600 ppm F) to all eligible dentin caries lesions on the contralateral side of the mouth. Single application per manufacturer's instructions.
  Interventions: Drug: Sodium Fluoride Varnish (5%)

INTERVENTIONS:
Drug: Sodium Fluoride Varnish (5%) — Topical application of 5% sodium fluoride varnish (22,600 ppm fluoride) to cavitated dentin caries lesions (ICDAS 3-5) on the contralateral side of the mouth. Applied once using a disposable applicator per manufacturer's instructions. This distinguishes it from lower-concentration fluoride gels or multiple-application protocols in other clinical trials.
  Arms: Fluoride Varnish (FV)
Drug: Silver Diamine Fluoride (38%) — Topical application of 38% silver diamine fluoride solution (44,800 ppm fluoride) to cavitated dentin caries lesions (ICDAS 3-5) on the assigned side of the mouth. Applied once with a microbrush for 1 minute, per manufacturer's instructions, without subsequent rinsing. This concentration and protocol distinguish it from other concentrations of SDF or repeated-application protocols used in other clinical studies."
  Arms: Silver Diamine Fluoride (SDF)

SUMMARY:
This randomized split-mouth clinical trial will compare the effectiveness of 38% silver diamine fluoride (SDF) versus 5% sodium fluoride varnish (FV) in reducing salivary Streptococcus mutans levels in children with bilateral caries. Each participant will receive SDF on one side of the mouth and FV on the contralateral side. The primary outcome is change in Dentocult SM Strip Mutans scores in plaque over 3 months. Secondary outcomes include plaque index, bleeding on probing, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-8 years; cooperative (Frankl ≥2).
* ≥2 contralateral primary molars with active dentin caries (ICDAS 3-5) of comparable severity.
* Parent/guardian consent; child assent when appropriate.

Exclusion Criteria:

* Silver allergy; ulcerative gingivitis/stomatitis.
* Systemic antibiotics within 4 weeks.
* Fixed appliances interfering with plaque assessment.
* Conditions precluding safe participation per clinician judgment.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Streptococcus mutans levels measured by Dentocult SM Strip Mutans test at baseline, 1 week, 1 month, and 3 months | 3 month
  Streptococcus mutans levels will be assessed using the Dentocult SM Strip Mutans test (Orion Diagnostica/Aidian). The test provides a semi-quantitative estimate of salivary S. mutans based on colony density on a selective culture strip.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No